CLINICAL TRIAL: NCT00658658
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Panitumumab in Children With Solid Tumors
Brief Title: Panitumumab in Children With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050252; 2014-005190-36 (EudraCT Number)
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Solid Tumors
Keywords: Epidermal Growth Factor; Pediatric; Solid Tumors; Panitumumab; Dose Limiting Toxicity
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): Participants received panitumumab at planned doses ranging from 2.5 mg/kg weekly (QW) to 9.0 mg/kg every 3 weeks (Q3W) until the patient experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
  Interventions: Biological: Panitumumab

INTERVENTIONS:
Biological: Panitumumab — Panitumumab administered by intravenous infusion
  Other Names: Vectibix

SUMMARY:
The primary objective of this study was to evaluate the safety and pharmacokinetics of up to 3 different dose schedules of panitumumab in pediatric patients with solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single arm, dose-ranging, clinical study. Panitumumab will be administered by intravenous infusion to 4-6 patients per cohort. Three planned cohorts, stratified by age, will be studied at 100% of the recommended panitumumab dose for each treatment schedule as defined in adults. Enrollment will start with a 2.5 mg/kg once weekly administration to the 12 to < 18 year old patients. Upon demonstration of sufficient safety additional cohorts will open; a 2.5 mg/kg once weekly administration to the 1 to < 12 year old patients and a 6.0 mg/kg once every two weeks to the 12 to < 18 year old patients. The decision to advance to the next cohort will be based on observance of ≤ 33% incidence of a dose limiting toxicity during the evaluation period. Subsequent cohorts of 6.0 mg/kg once every two weeks to the 1 to < 12 year old patients and 9.0 mg/kg once every three weeks to both age groups will open once sufficient safety in each cohort is determined. Participants may stay on study treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardian signed-written informed consent
* 1 to < 18 years of age
* Histologically or cytologically confirmed solid tumor that has recurred after standard therapy, or for which there is no standard therapy. Subjects with brainstem glioma DO NOT need histologic proof of the diagnosis.
* Paraffin-embedded tumor tissue from primary tumor or metastasis for determination of epidermal growth factor receptor expression and biomarker testing
* Central nervous system tumors are allowed
* Presence of measurable or non-measurable disease.
* Life expectancy of ≥ 12 weeks.
* Performance status: Karnofsky ≥ 60% for 12 to <18 years of age; Lansky play scale ≥ 60% for 1 to < 12 years of age.
* Adequate hematologic function.
* Adequate renal function.
* Adequate hepatic function.
* Magnesium ≥ lower limit of normal (LLN)
* Adequate pulmonary function
* All previous therapy-related toxicities must have resolved or return to baseline.

Exclusion Criteria:

* Diagnosis of leukemia, non-Hodgkin's lymphoma, Hodgkin's disease or other hematologic malignancy.
* Any prior allogeneic transplant.
* Prior autologous bone marrow or peripheral stem cell transplant less than 3 months prior to enrollment.
* Substantial radiotherapy to the bone marrow within 6 weeks prior to enrollment.
* Prior use of any monoclonal antibodies directly targeting the epidermal growth factor receptor (EGFr). Subjects who have received prior tyrosine kinase inhibitors such as gefitinib or erlotinib are eligible.
* Immunotherapy, radiotherapy, or chemotherapy ≤ 2 weeks prior to enrollment. (≤ 6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin, and ≤ 6 weeks from prior antibody therapy).
* Requirement to receive concurrent chemotherapy, immunotherapy, radiotherapy (except for pain control) or any other investigational drug while on this study.
* Prior seizures < 3 months prior to enrollment. Subjects with a history of seizure disorders ≥ 3 months prior to enrollment must be seizure free and on stable anticonvulsant medication(s) for ≥ 3 months prior to enrollment).
* Presence of a serious uncontrolled medical disorder.
* Dementia, altered mental status, or any other medical condition or disorder that would prohibit the understanding or rendering of assent (if applicable), or ability to comply with study procedures.
* Major surgery ≤ 28 days prior to enrollment.
* Known or suspected history of interstitial lung disease.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea.
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, acute or chronic hepatitis B infection, or any co-morbid disease that would increase risk of toxicity.
* Females of childbearing potential not using adequate contraception precautions for the duration of the study treatment and for 2 months after the last administration of investigational product.
* Pregnant or breast-feeding, or planning to become pregnant during study treatment and within 2 months after the last administration of investigational product.
* Received investigational therapy or procedure ≤ 30 days prior to enrollment.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (11):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Minneapolis, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in the United States. Participants were enrolled from 14 March 2008 to 4 March 2015.
Pre-assignment Details: Three dose regimens were to be tested in pediatric patients stratified by age group (1 to 11 versus 12 to 17 years). Participants were enrolled sequentially into each dose group, beginning with the 2.5 mg/kg, 12 to 17 year old cohort, based upon demonstration of sufficient safety.
Groups:
- Age 12-17: 2.5 mg/kg QW: Participants aged 12 to 17 years received panitumumab 2.5 mg/kg administered by intravenous (IV) infusion weekly (QW) until the participant experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
- Age 12-17: 6 mg/kg Q2W: Participants aged 12 to 17 years received panitumumab 6 mg/kg administered by IV infusion every 2 weeks (Q2W) until the participant experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
- Age 12-17: 9 mg/kg Q3W: Participants aged 12 to 17 years received panitumumab 9 mg/kg administered by IV infusion every 3 weeks (Q3W) until the participant experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
- Age 1-11: 2.5 mg/kg QW: Participants aged 1 to 11 years received panitumumab 2.5 mg/kg administered by IV infusion QW until the participant experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
- Age 1-11: 6 mg/kg Q2W: Participants aged 1 to 11 years received panitumumab 6 mg/kg administered by IV infusion Q2W until the participant experienced disease progression, was unable to tolerate study drug, withdrew consent, or other reasons that warranted removal from the study.
Period: Overall Study
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Started | 6 | 7 | 4 | 6 | 8
Completed | 1 | 5 | 4 | 4 | 3
Not Completed | 5 | 2 | 0 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Death | 4 | 0 | 0 | 1 | 1
Not completed — Disease Progression | 0 | 1 | 0 | 1 | 3
Not completed — Protocol-specified Criteria | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W | Total
Number analyzed (Participants) | 6 | 7 | 4 | 6 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (0.8) | 15.6 (1.5) | 15.8 (1.9) | 7.8 (3.1) | 8.4 (2.8) | 11.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 3 | 4 | 14
  Male | 3 | 6 | 1 | 3 | 4 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Black (or African American) | 1 | 1 | 0 | 1 | 0 | 3
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 2
  Other | 0 | 0 | 0 | 1 | 0 | 1
  White or Caucasian | 5 | 4 | 3 | 4 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: Any panitumumab related grade 3 or 4 hematologic or non-hematologic toxicity (graded according to the modified Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 criteria) was considered a DLT with the exception of alopecia and fatigue. Hypomagnesemia, nausea, diarrhea, vomiting, and skin or nail toxicities constituted a DLT only of the following occured: • Grade 3 or 4 hypomagnesemia that persisted for at least 5 days despite maximal magnesium replacement; • Grade 3 or 4 diarrhea, nausea, or vomiting that persisted for at least 5 days despite maximum supportive therapy; • Grade 4 skin or nail toxicity.
Time Frame: 28 days from initial administration of panitumumab for the 2.5 and 6 mg/kg cohorts and 21 days from first administration for the 9 mg/kg cohort.
Population: DLT Analysis Set (all participants who received at least 1 dose of panitumumab and were evaluated for DLTs and completed at least 28 days (for the 2.5 and 6 mg/kg cohorts) or 21 days (for 9 mg/kg cohort) of therapy unless due to a DLT)
Measure: Number; unit: participants
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 5
participants | 1 | 0 | 0 | 1 | 3

2. Secondary Outcome: Number of Participants Who Developed Antibodies to Panitumumab
Description: Three validated assays were used to detect the presence of anti-panitumumab antibodies. Two screening immunoassays, an acid-dissociation enzyme-linked immunosorbent assay (ELISA) and a Biacore-based biosensor assay, were used to detect antibodies capable of binding to panitumumab. All samples confirmed to be positive by drug specificity in either screening immunoassay were further tested for neutralizing antibodies in a cell-based epidermal growth factor receptor (EGFR) phosphorylation bioassay. The number of participants who developed antibodies to panitumumab is the number of participants with a non-positive (including missing) antibody result at baseline and a positive antibody result at any post-baseline time point.
Time Frame: Before panitumumab administration on Day 1, Day 43, Day 169 and 30 days after last dose for all cohorts.
Population: Safety Analysis Set participants with at least one post-baseline immunoassay result
Measure: Number; unit: participants
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 5 | 4 | 3 | 4
participants
  Binding antibodies | 1 | 0 | 0 | 2 | 0
  Neutralizing antibodies | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event is defined as an AE that: • is fatal; • is life threatening; • requires in-patient hospitalization or prolongation of existing hospitalization; • results in persistent or significant disability/incapacity; • is a congenital anomaly/birth defect; • other significant medical hazard. The investigator assessed whether adverse events were related to panitumumab. The severity of adverse events was based on CTCAE version 3 (with the exception of skin- or nail-related toxicities which were graded using the CTCAE version 3.0 with modifications), according to the following: Grade 1 = Mild (aware of sign or symptom, but easily tolerated); Grade 2 = Moderate (discomfort enough to cause interference with usual activity); Grade 3 = Severe (incapacitating with inability to work or do usual activity); Grade 4 = Life-threatening or disabling; Grade 5 = Fatal.
Time Frame: From first dose date to end of study date. The median duration of study was 47 days.
Population: Safety Analysis Set (all participants who received at least 1 dose of panitumumab)
Measure: Number; unit: participants
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 6 | 7 | 4 | 6 | 8
participants
  Any adverse event | 6 | 7 | 3 | 6 | 8
  Serious adverse events | 5 | 3 | 2 | 3 | 5
  Treatment-related adverse event | 5 | 5 | 3 | 5 | 6
  Treatment-related serious adverse event | 1 | 0 | 0 | 1 | 2
  Withdrawals due to adverse event | 0 | 0 | 0 | 0 | 0
  Grade 1 | 5 | 7 | 3 | 6 | 6
  Grade 2 | 5 | 6 | 3 | 4 | 7
  Grade 3 | 4 | 5 | 2 | 4 | 6
  Grade 4 | 4 | 0 | 0 | 1 | 2
  Fatal | 4 | 0 | 0 | 1 | 1

4. Primary Outcome: Maximum Observed Concentration (Cmax) of Panitumumab
Description: Panitumumab serum concentration was measured using an enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) of the assay was 400 pg/mL. Concentrations below the LLOQ were set to zero.
Time Frame: First dose (Day 1) and third dose (Day 15/29/43 for the QW, Q2W and Q3W cohorts respectively). Samples were collected over the dosing interval for each treatment cohort (7, 14 or 21 days for QW, Q2W and Q3W cohorts respectively).
Population: Pharmacokinetic (PK) Analysis Set (all participants who received the correct dose of panitumumab and from whom the PK parameters could be assessed); "n" indicates the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 6 | 7 | 3 | 4 | 7
μg/mL
  First Dose (n=6, 7, 3, 4, 7) | 52.8 (11.4) | 161 (41.2) | 205 (45.9) | 42.9 (8.51) | 120 (29.4)
  Third Dose (n=3, 5, 1, 3, 2) | 76.6 (21.1) | 187 (45.2) | 327 (NA) — Cannot be calculated when n = 1 | 60.8 (15.7) | 126 (NA) — Not calculated as not considered reliable when n = 2

5. Primary Outcome: Minimum Observed Concentration (Cmin) of Panitumumab
Time Frame: as for outcome 4
Population: PK analysis set; "n" indicates the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 7 | 2 | 4 | 5
μg/mL
  First Dose (n=4, 7, 2, 4, 5) | 6.62 (6.83) | 24.7 (18.6) | 35.3 (NA) — Not calculated as not considered reliable when n = 2 | 4.87 (3.64) | 19.7 (15.5)
  Third Dose (n=3, 5, 0, 3, 2) | 24.2 (22.9) | 48.1 (25.1) | NA (NA) — No participants with available data | 17.3 (8.83) | 26.1 (NA) — Not calculated as not considered reliable when n = 2

6. Primary Outcome: Area Under the Concentration-time Curve During the Dosing Interval (AUC0-tau) for Panitumumab
Description: The area under the serum concentration-time curve from time zero to the end of the dosing interval (AUCtau), estimated using the linear trapezoidal method.
Time Frame: as for outcome 4
Population: PK analysis set; "n" indicates the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 7 | 2 | 4 | 5
day*μg/mL
  First Dose (n=4, 7, 2, 4, 5) | 167 (86.1) | 1040 (357) | 1580 (NA) — Not calculated as not considered reliable when n = 2 | 127 (37.9) | 708 (247)
  Third Dose (n=3, 5, 0, 3, 2) | 306 (178) | 1330 (357) | NA (NA) — No participants with available data | 255 (70.7) | 754 (NA) — Not calculated as not considered reliable when n = 2

7. Primary Outcome: Half-life (t1/2) for the Terminal Phase (First Dose) or Dosing Interval (Third Dose) of Panitumumab
Time Frame: as for outcome 4
Population: PK analysis set; "n" indicates the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 2 | 5 | 1 | 3 | 3
days
  First Dose (n=2, 5, 1, 3, 3) | 1.33 (NA) — Not calculated as not considered reliable when n = 2 | 4.49 (1.09) | 4.27 (NA) — Cannot be calculated when n = 1 | 2.11 (0.913) | 4.23 (1.64)
  Third Dose (n=2, 2, 0, 1, 1) | 2.94 (NA) — Not calculated as not considered reliable when n = 2 | 4.98 (NA) — Not calculated as not considered reliable when n = 2 | NA (NA) — No participants with available data | 3.07 (NA) — Cannot be calculated when n = 1 | 4.91 (NA) — Cannot be calculated when n = 1

8. Primary Outcome: Serum Clearance (CL) of Panitumumab
Time Frame: as for outcome 4
Population: PK analysis set; "n" indicates the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 3 | 5 | 1 | 4 | 3
mL/day/kg
  First Dose (n=3, 5, 1, 4, 3) | 19.8 (8.57) | 6.38 (0.466) | 7.15 (NA) — Cannot be calculated when n = 1 | 18.7 (6.35) | 8.06 (1.40)
  Third Dose (n=3, 5, 0, 3, 2) | 9.92 (4.40) | 4.69 (1.00) | NA (NA) — No participants with available data | 10.1 (2.44) | 8.05 (NA) — Not calculated as not considered reliable when n = 2

9. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Disease assessments were based on investigator review of scans using modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 criteria. A participant was considered a responder if their best response was either a complete or partial response. Participants without a post-baseline assessment were considered non-responders. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met. Complete Response (CR): Disappearance of all target and non-target lesions, normalization of tumor markers and no new lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions, no progression of non-target lesions and no new lesions, or, the disappearance of all target lesions, persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease (PD) or/and maintenance of tumor marker level above normal limits, and no new lesions.
Time Frame: Tumor response was assessed every 8 weeks through week 48 and every 3 months thereafter until disease progression or end of study. The data cut-off for the analysis was 17 June 2015; median duration of study was 47 days.
Population: Safety Analysis Set participants with presence of baseline measurable disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 3 | 4 | 2 | 3
percentage of participants | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 70.76]

10. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease assessments were based on investigator review of scans using modified RECIST version 1.0 criteria. A participant was considered to have disease control if their best response is either a complete or partial response, or stable disease. Participants without a post-baseline assessment were considered to not have disease control. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met. A best overall response of SD requires a visit response of SD or better, no earlier than 49 days after the date of enrollment.
  Stable disease (SD): Neither sufficient shrinkage of target lesions to qualify for a PR nor sufficient increase to qualify for PD and no progression of existing non-target lesions and no new lesions.
Time Frame: as for outcome 9
Population: Safety Analysis Set participants with presence of baseline measurable disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Number analyzed (Participants) | 4 | 3 | 4 | 2 | 3
percentage of participants | 0.00 [0.00 to 60.24] | 33.33 [0.84 to 90.57] | 0.00 [0.00 to 60.24] | 50.00 [1.26 to 98.74] | 66.67 [9.43 to 99.16]

ADVERSE EVENTS:
Time Frame: From first dose date to end of study date. The median duration of study is 47 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those participants who received at least one dose of investigational product.
Arm/Group | Age 12-17: 2.5 mg/kg QW | Age 12-17: 6 mg/kg Q2W | Age 12-17: 9 mg/kg Q3W | Age 1-11: 2.5 mg/kg QW | Age 1-11: 6 mg/kg Q2W
Serious Adverse Events (participants affected / at risk) | 5/6 | 3/7 | 2/4 | 3/6 | 5/8
Other Adverse Events (participants affected / at risk) | 5/6 | 7/7 | 3/4 | 6/6 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age 12-17: 2.5 mg/kg QW (N=6) | Age 12-17: 6 mg/kg Q2W (N=7) | Age 12-17: 9 mg/kg Q3W (N=4) | Age 1-11: 2.5 mg/kg QW (N=6) | Age 1-11: 6 mg/kg Q2W (N=8)
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age 12-17: 2.5 mg/kg QW (N=6) | Age 12-17: 6 mg/kg Q2W (N=7) | Age 12-17: 9 mg/kg Q3W (N=4) | Age 1-11: 2.5 mg/kg QW (N=6) | Age 1-11: 6 mg/kg Q2W (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 4 | 2 | 0 | 2
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Temperature difference of extremities (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Bone atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 2
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Phantom pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.